CLINICAL TRIAL: NCT05060822
Title: A Phase II, Multi-center, Randomized, Placebo-controlled (Double-blind Design), Active Comparator-controlled (Open-label Design), Parallel-group, Dose-finding Study, to Evaluate the Efficacy and Safety of HEC585 Tablets in Patients With IPF
Brief Title: Phase ll Study of HEC585 in Patients With IPF
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sunshine Lake Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HEC585-P-03
Record Dates: First submitted 2021-09-18; First posted 2021-09-29 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-04

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — pirfenidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: placebo-controlled (double-blind design), active comparator-controlled (open-label design)，parallel-group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- HEC585 dose A (Experimental): Drug: HEC585 dose A once daily, up to 24 weeks-120 weeks
  Interventions: Drug: HEC585
- HEC585 dose B (Experimental): Drug: HEC585 dose B once daily, up to 24 weeks-120 weeks
  Interventions: Drug: HEC585
- HEC585 dose C (Experimental): Drug: HEC585 dose C once daily, up to 24 weeks-120 weeks
  Interventions: Drug: HEC585
- pirfenidone (Active Comparator): Drug: pirfenidone three times a day (target dose), up to 24 weeks
  Interventions: Drug: Pirfenidone
- placebo (Placebo Comparator): Drug: placebo once daily, up to 24 weeks-120 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HEC585 — HEC585 Tablets，once daily
  Arms: HEC585 dose A; HEC585 dose B; HEC585 dose C
Drug: Pirfenidone — Pirfenidone，three times a day
  Arms: pirfenidone
Drug: Placebo — Placebo，once daily
  Arms: placebo

SUMMARY:
A Phase ll Study to evaluate the efficacy and safety of various doses of HEC585 Tablets in patients with idiopathic pulmonary fibrosis

ELIGIBILITY:
Inclusion Criteria:

* Volunteer to participate in this clinical study and sign the ICF before the study begins;
* Aged 40-80 (including 40 and 80) ;
* Female or male subjects with child-bearing potential who agree and promise to take effective contraceptive measures;
* Diagnosed with IPF according to the Official ATS/ERS/JRS/ALAT Clinical Practice Guideline for IPF Diagnosis (2018);
* FEV1/FVC ≥ 0.7;
* FVC ≥ 45% predicted;
* DLCO corrected for Haemoglobin (Hb) ≥ 30% predicted of normal;
* In the opinion of the Investigator, subjects are willing and able to comply with the protocol requirements and attend the visit.

Exclusion Criteria:

* In the opinion of the Investigator, subjects underwent significant deterioration in IPF within one month before randomization;
* Interstitial lung disease caused by other known causes;
* Any bacterial, viral, parasitic or fungal infection that needs to be treated at screening;
* Expected to receive lung transplantation during the study;
* Expected survival is less than 6 months;
* History of tumors within 5 years before screening (except for localized cancers such as basal cell carcinoma);
* Moderate to severe hepatic insufficiency (Child-Pugh grade B or C, see Appendix 4);
* History of unstable or worsening heart disease within 6 months before screening;
* Cannot perform 6MWT or PFT;
* Allergic to any component of HEC585 Tablets or pirfenidone tablets;
* Participated in other clinical study and received the last dose within 3 months before screening;
* Pregnant or breastfeeding;
* History of smoking within 3 months before screening or are unwilling to quit smoking during the study;
* Subjects often drink alcohol within 6 months before the screening (drink more than 21 units of alcohol a week), or refuse to reduce alcohol intake during the study;
* History of drug abuse within 6 months before the screening;
* Family or personal history of QT prolongation syndrome;
* Any condition that, in the opinion of the investigator, would compromise the safety or compliance of the subject, or prevent the subject from completing the study.
* TBil > 1.5 × ULN or AST or ALT > 2 × ULN;
* CLcr < 50 mL/min;
* Human immunodeficiency virus (HIV) antibody is positive;
* Uncontrolled hepatitis B virus infection or hepatitis C virus infection;
* QTcF > 480 ms.
* Subjects have received any of the following treatments within 28 days before randomization:

  1. Any cytotoxic drug or immunosuppressant
  2. Therapeutic drugs for IPF, including but not limited to pirfenidone, nintedanib, prednisone at > 15 mg/d or other glucocorticoids of the equivalent dose, N-acetylcysteine at > 600 mg/d.
  3. Moderate and strong inhibitor or strong inducer of CYP1A2.
  4. Strong inducers or strong CYP3A4 inhibitors.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2021-06-30 (Actual); Primary Completion 2024-05-10 (Estimated); Study Completion 2025-05-11 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline to Week 24 in %FVC compared with placebo | 24 Weeks
  change in %FVC, measured using Spirometer, from baseline to week 24

SECONDARY OUTCOMES:
Change from Baseline to Week 24 in %FVC compared with Pirfenidone | 24 Weeks
  change in %FVC, measured using Spirometer, from baseline to week 24
Change from Baseline to Week 12 in %FVC compared with placebo/ Pirfenidone | 12 Weeks
  change in %FVC, measured using Spirometer, from baseline to week 12
Proportion of subjects with an absolute decline from baseline in FVC (% predicted) of > 10% | 24 Weeks
  The proportion of subjects whose %FVC decline from baseline by more than 10% in each treatment group at W24
Time to first acute IPF exacerbation | 24 Weeks
All-cause mortality | 24 Weeks
IPF related mortality | 24 Weeks
Changes of 6MWT results | 12 Weeks, 24 Weeks
Changes of SGRQ scores | 12 Weeks, 24 Weeks
Changes of DLco (Hb correction) | 12 Weeks, 24 Weeks
Changes of resting SpO2 | 12 Weeks, 24 Weeks

CONTACTS AND LOCATIONS:
Locations (1):
- China-Japan Friendship Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No